CLINICAL TRIAL: NCT04544007
Title: A Phase II Trial of Poly-ICLC for Progressive, Previously Treated Low-Grade Gliomas in Children and Young Adults With Neurofibromatosis Type 1
Brief Title: A Phase II Trial of Poly-ICLC for Low-Grade Gliomas
Acronym: NF111
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The closure of the study is due to the lack of enrollment and the lack of evaluable patients.
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Children's Healthcare of Atlanta (Other); Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Bruce Korf, MD, Associate Dean for Genomic Medicine, UAB School of Medicine and Chief Genomics Officer, UAB Medicine, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W81XWH-17-2-0037
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: NF1; Low-grade Glioma
MeSH Terms: interventions — poly ICLC

STUDY DESIGN:
Intervention Model Description: Patients must be less than 22 years of age with a diagnosis of NF1 and LGG of the brain and spinal cord (WHO Grade 1 and 2)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administer Poly-ICLC (Experimental): Enrolled participants will receive poly-ICLC 20 mcg/kg/dose twice weekly IM (using Monday/Thursday or Tuesday/Friday schedule if possible).
  Interventions: Drug: Poly ICLC

INTERVENTIONS:
Drug: Poly ICLC — Enrolled participants will receive poly-ICLC 20 mcg/kg/dose twice weekly IM (using Monday/Thursday or Tuesday/Friday schedule if possible).
  Other Names: Hiltonol

SUMMARY:
This is a phase II, prospective, longitudinal, multi-center trial of poly-ICLC (Hiltonol ®) treatment for progressive low-grade gliomas in pediatric patients with NF1. The primary objective is to evaluate the efficacy of poly-ICLC in pediatric NF1 patients with progressive low-grade glioma (LGG) as measured by objective tumor response rate (CR+PR) within the first 48 weeks (12 cycles) of therapy. There will also be secondary and exploratory objectives listed in the detailed description below.

DETAILED DESCRIPTION:
This is a phase II, prospective, longitudinal, multi-center trial of poly-ICLC (Hiltonol ®) treatment for progressive low-grade gliomas in pediatric patients with NF1. The primary objective is to evaluate the efficacy of poly-ICLC in pediatric NF1 patients with progressive low-grade glioma (LGG) as measured by objective tumor response rate (CR+PR) within the first 48 weeks (12 cycles) of therapy.

The secondary objectives are to:

1. Determine 12, 24 and 60 month progression free survival (PFS) in pediatric NF1 patients with progressive LGG treated with poly-ICLC.
2. Evaluate the efficacy of poly-ICLC in pediatric NF1 patients with progressive LGG as measured by best objective tumor response rate (CR+PR) within 24 cycles of therapy.
3. Evaluate the efficacy of poly-ICLC in pediatric NF1 patients with progressive LGG as measured by clinical benefit response rate (CR+PR+MR+SD) after 12 and 24 cycles of therapy.
4. Assess the toxicity associated with poly-ICLC treatment in pediatric NF1 patients with LGG.

Exploratory objectives are to:

1. Evaluate the visual outcome measures in children with progressive optic pathway gliomas treated with poly-ICLC. Visual response is defined as 0.2 logMAR or greater in acuity improvement.
2. Evaluate patient reported outcomes and quality of life measures.
3. Evaluate biological correlates.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Patients must be less than 22 years at the time of enrollment; there is no lower age limit.
2. All participants must have an identified pathogenetic constitutional NF1 mutation OR the clinical diagnosis of NF1 using the NIH Consensus Conference criteria.
3. Diagnosis: LGG (WHO Grade 1 and 2) of the brain and spinal cord are eligible. Histologic confirmation of tumor is not necessary in the presence of consistent clinical and radiographic findings. Biopsy for histologic diagnosis is required if there is clinical suspicion for a high-grade tumor; special attention is recommended in older adolescents or young adults to the potential for malignant transformation. Patients with metastatic disease are eligible.
4. Patients must meet at least one of the following criteria for progression or recurrence of a previously treated target tumor:

   1. Progression or recurrence on MRI.
   2. New or worsening neurologic symptoms attributable to the target tumor.
   3. For patients with OPG: visual worsening, defined as worsening of visual acuity (VA) or visual fields (VF) documented within the past year by examination or history, attributable to tumor.
5. Measurable Disease: Patients must have two-dimensional measurable tumor >1cm2.
6. Prior Therapy: Patients must have had at least one prior medical treatment for the target LGG.
7. Performance Level: Patients must have a performance status of equal or > than 50 using Karnofsky for patients equal or ≥ 16 years of age and Lansky for patients < 16 years of age.
8. Patients must have recovered to grade ≤1 from any acute toxicities from all prior treatments. to enroll on this study and meet time restrictions from end of prior therapy as defined below:

   1. Myelosuppressive chemotherapy: must have received the last dose of myelosuppressive therapy at least 4 weeks prior to study registration, or at least 6 weeks if nitrosourea.
   2. Investigational/biological agent: Patient must have received the last dose of other investigational, immunotherapy, or biological agent > 14 days prior to study registration or at least 5 half-lives, whichever is greater. Bevacizumab last dose > 36 days prior to enrollment.
   3. Radiation therapy: Patients SHOULD NOT have received prior irradiation.
   4. Study specific limitations on prior therapy: There is no limit on the number of prior treatment regimens.
   5. Growth factor(s): Must not have received any hematopoietic growth factors within 7 days of study entry or > 14 days if pegylated GCSF is used.
   6. Prior surgery: At the time of enrollment, must be ≥ 3 weeks from prior major surgery such as craniotomy, orthopedic surgery, abdominal surgery or ≥1 week from minor surgery and completely recovered. Port or central line placement is not considered a major surgery.
9. Organ Function Requirements:

   All patients must have adequate organ function defined as:

   9.1 Hematologic Function:
   1. Hemoglobin: > 8.0 gm/dl (may transfuse PRBCs)
   2. ANC: > 750/mm3. Must be at least 7 days after last dose of growth factor or > 14 days since last dose of pegylated GCSF
   3. Platelet Count: > 75,000/mm3 (transfusion independent; ≥ 7 days from last transfusion)

   9.2 Renal Function: Serum creatinine which is less than 1.5 times ULN for age (as per the table below) or GFR > 70 ml/min/1.73m2

   Renal Function Normal for Age

   Age Maximum Serum Creatinine (mg/dL) Male Female 1 month to < 6 months 0.4 0.4 6 months to < 1 year 0.5 0.5 1 to < 2 years 0.6 0.6 2 to < 6 years 0.8 0.8 6 to < 10 years 1 1 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.4

   ≥ 16 years 1.7 1.4

   Liver Function:
   1. Total bilirubin < 1.5 x ULN (Children with diagnosis of Gilbert's Syndrome will be allowed on the study regardless of their total and indirect bilirubin levels as long as the direct bilirubin is less than 3.1 mg/dL.)
   2. SGPT (ALT) ≤ 5 x ULN
   3. SGOT (AST) ≤ 5 x ULN

   Pulmonary Function:

   No evidence of dyspnea at rest, and a pulse oximetry ≥ 92%.

   Reproductive Function:

   Female patients of childbearing potential must have negative serum or urine pregnancy test within 7 days prior to the first dose of poly-ICLC. Patient must not be pregnant or breast-feeding. Patients of childbearing or child-fathering potential must be willing to use a medically acceptable form of birth control, including abstinence, while being treated on this study and for 90 days following cessation of treatment.
10. Patient is able to start treatment within 7 days after enrollment.
11. Patients with neurological deficits must be stable for a minimum of 1 week prior to enrollment.
12. Patients are only eligible if complete resection of the LGG with acceptable morbidity is not feasible, or if a patient with a surgical option refuses surgery.
13. Parents/legal guardians must provide written informed consent and agree that they will comply with the study.

Exclusion Criteria:

1. Prior radiation treatment for the low-grade glioma.
2. Prior exposure to poly-ICLC.
3. Patients currently receiving other anti-tumor therapy or experimental therapy (targeted agents, chemotherapy radiation).
4. Patients with a current or prior diagnosis of malignant glioma (WHO grade III or IV).
5. Patients with a prior diagnosis of malignant peripheral nerve sheath tumor or other malignancy requiring treatment in the last 48 months.
6. Patients may not have fever (≥38.50 C) within 3 days of enrollment.
7. Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.
8. Active auto-immune illness.
9. Pregnant or lactating females.
10. Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation and for 90 days after stopping study therapy are not eligible.
11. Severe unresolved infection that requires systemic IV antibiotics.
12. Patients with any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy.
13. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, impaired gastrointestinal function, or psychiatric illness/social situations that would limit compliance with study requirements.
14. Patients requiring high doses of steroids. Patients may not be on immunosuppressive therapy, including corticosteroids (with the exception of physiologic replacement, defined as ≤ 0.75 mg/m2/day dexamethasone or equivalent) at time of enrollment. However, patients who require intermittent use of bronchodilators or local steroid injections will not be excluded from the study.

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juliette Southworth, BS, CCRP, Study Director — University of Alabama at Birmingham, NFCTC
Locations (12):
- United States (12):
  - The University of Alabama at Birmingham (Site 700), Birmingham, Alabama
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's National Medical Center (Site 775), Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Children's Lurie Hospital, Chicago, Illinois
  - Lurie Children's Hospital of Chicago (Site 350), Chicago, Illinois
  - University of Chicago (Site 850), Chicago, Illinois
  - Washington University - St. Louis (Site 900), St Louis, Missouri
  - New York University Medical Center (Site 200), New York, New York
  - Cincinnati Children's Hospital Medical Center (Site 800), Cincinnati, Ohio
  - Children's Hospital of Philadelphia (Site 750), Philadelphia, Pennsylvania
  - Childrens Medical Center - Univ. of Texas SW (Site 917), Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Administer Poly-ICLC
Started | 3
Completed | 1
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Confirmed Progressive Disease | 1

BASELINE CHARACTERISTICS:
Population: Participants will receive therapy with poly-ICLC at a dose of 20 mcg/kg/dose IM injections twice a week up to 24 cycles (a cycle consists of 28 days) from the start of poly-ICLC in the absence of disease progression or significant toxicity.
Groups:
- Poly-ICLC: This is a phase II, prospective, longitudinal, multi-center trial of poly-ICLC (Hiltonol) treatment for progressive low-grade gliomas in pediatric patients with NF1. The primary objective is to evaluate the efficacy of poly-ICLC in pediatric NF1 patients with progressive low-grade glioma (LGG) as measured by objective tumor response rate (CR+PR) within the first 48 weeks (12 cycles) of therapy.
Arm/Group | Poly-ICLC
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11 (6.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3
Poly-ICLC [Count of Participants; unit: Participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Efficacy of Poly-ICLC
Description: Evaluate the efficacy of poly-ICLC in pediatric NF1 patients with progressive low-grade glioma (LGG) as measured by objective tumor response rate (CR+PR), using Response Assessment in Pediatric Neuro-Oncology (RAPNO) criteria. Complete Response (CR) is complete disappearance of the target lesion on T2 weighted and T2 weighted fluid attenuated inversion recovery (FLAIR) imaging and contrast imaging using baseline MRI or best recorded response for comparison; Partial Response (PR) is 50% or greater reduction in the target lesion on T2 weighted and T2 weighted-FLAIR imaging using the baseline MRI for comparison. Response will be assessed through the time of the post-12th cycle tumor assessment, or through the last tumor assessment time during this nominal period for patients in follow-up but who have withdrawn from protocol therapy, or through the last available tumor assessment for patients who are lost to follow-up during this time.
Time Frame: First 48 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Poly-ICLC: Enrolled participants will receive poly-ICLC 20 mcg/kg/dose twice weekly IM
Arm/Group | Poly-ICLC
Number analyzed (Participants) | 3
Participants
  Achieved Complete or Partial Response | 0
  Failed to Achieve Complete or Partial Response | 3

2. Secondary Outcome: Determine Progression Free Survival (PFS)
Description: Determine progression free survival (PFS) in pediatric NF1 patients with progressive LGG treated with poly-ICLC. Progression free survival (PFS), defined as the time from start of treatment to the first occurrence of tumor recurrence, tumor progression, occurrence of a second malignancy, or death from any cause. Patients event-free at last follow-up will be censored in analysis. PFS will be determined at 12, 24 and 60 months.
Time Frame: 12 months
Population: 1 patient progressed on day 170. The other 2 patients are censored on day 134 and day 849 respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Poly-ICLC
Number analyzed (Participants) | 3
Participants
  Progressed by last visit | 1
  Censored at the last visit | 2

3. Secondary Outcome: Determine Progression Free Survival (PFS)
Description: as for outcome 2
Time Frame: 24 Months
Population: 1 patient progressed on day 170. The other 2 patients are censored on day 134 and day 849 respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Administer Poly-ICLC
Number analyzed (Participants) | 3
Participants
  Progressed by last visit | 1
  Censored at the last visit | 2

4. Secondary Outcome: Number of Participants Who Achieved Best Objective Tumor Response Rate (CR+PR)
Description: Evaluate the efficacy of poly-ICLC in pediatric NF1 patients with progressive LGG as measured by best objective tumor response rate (CR+PR) within 24 cycles of therapy. Objective response rate (defined as CR or PR) after 24 cycles of treatment. Response will be assessed through the time of the post-24th cycle tumor assessment, or through the last tumor assessment time during this nominal period for patients in follow-up, but who have withdrawn from protocol therapy, or through the last available tumor assessment for patients who are lost to follow-up during this time.
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Administer Poly-ICLC
Number analyzed (Participants) | 3
Participants
  Achieved Complete or Partial Response | 0
  Failed to Achieve Complete or Partial Response | 3

5. Secondary Outcome: Evaluate Efficacy by Clinical Benefit Response Rate (CR+PR+MR+SD)
Description: Evaluate the efficacy of poly-ICLC in pediatric NF1 patients with progressive LGG as measured by clinical benefit response rate (CR+PR+MR+SD). Clinical benefit defined as (CR+PR+MR+SD). Clinical benefit will be assessed through the time of the post-12 and 24th cycle tumor assessment, or through the last tumor assessment time during this nominal period for patients in follow-up but who have withdrawn from protocol therapy, or through the last available tumor assessment for patients who are lost to follow-up during this time.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Poly-ICLC
Number analyzed (Participants) | 3
Participants
  Complete Response at 12 Months | 0
  Partial Response at 12 Months | 0
  Minor Response at 12 Months | 0
  Stable Disease at 12 Months | 1
  Progressive Disease at 12 Months | 1
  Failed to Remain on Treatment for 12 Months | 1

6. Secondary Outcome: Evaluate Efficacy by Clinical Benefit Response Rate (CR+PR+MR+SD)
Description: as for outcome 5
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Poly-ICLC
Number analyzed (Participants) | 3
Participants
  Complete Response at 24 Months | 0
  Partial Response at 24 Months | 0
  Minor Response at 24 Months | 0
  Stable Disease at 24 Months | 1
  Progressive Disease at 24 Months | 0
  Failed to reach at 24 Months | 2

7. Secondary Outcome: Assess Toxicity
Description: Assess the toxicity associated with poly-ICLC treatment in pediatric NF1 patients with LGG. The grade and duration of CTCAE toxicities observed during treatment, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Event (CTCAE) version 5.0 for reporting of adverse events.
Time Frame: Up to 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Poly-ICLC
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: Up to 24 Months
Description: Assess the toxicity associated with poly-ICLC treatment in pediatric NF1 patients with LGG
Groups:
- Poly-ICLC: This is a phase II, prospective, longitudinal, multi-center trial of poly-ICLC (Hiltonol) treatment for progressive low-grade gliomas in pediatric patients with NF1. The primary objective is to evaluate the efficay of poly-ICLC in pediatric NF1 patients with progressive low-grade glioma (LGG) as measured by objective tumor response rate (CR+PR) within the first 48 weeks (12 cycles) of therapy.
Arm/Group | Poly-ICLC
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Poly-ICLC (N=3)
Middle Ear Inflammation (Ear and labyrinth disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Poly-ICLC (N=3)
White Blood Cell Decreased (Blood and lymphatic system disorders) | 1 (1)
Middle Ear Inflammation (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Eye Disorders - Other, Proptosis (Eye disorders) | 1 (1)
Periorbital Edema (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Injection Site Reaction (General disorders) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Otitis Media (Infections and infestations) | 1 (2)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Neutrophil Count Decreased (Investigations) | 1 (1)
Weight Gain (Investigations) | 1 (2)
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 (11)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and Connective Tissue Disorder - Other, Specify, Joint Crepitus (Musculoskeletal and connective tissue disorders) | 1 (1)
Facial Muscle Weakness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (5)
Hydrocephalus (Nervous system disorders) | 1 (3)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT04544007/Prot_SAP_003.pdf
  • Informed Consent Form (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT04544007/ICF_002.pdf